CLINICAL TRIAL: NCT03507348
Title: Evaluation of Desensitization Protocols in HLA-incompatible Kidney-transplant Candidates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigateur decision
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC17.247
Record Dates: First submitted 2018-03-23; First posted 2018-04-25 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: End-stage Renal Disease; Kidney Transplantation; Hla-incompatible Kidney Transplant Candidates
Keywords: Anti-HLA alloantibodies; Desensitization therapy; Tocilizumab; Rituximab
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Rituximab; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desensitization with Tocilizumab and rituximab (MFI >15000) (Other)
  Interventions: Drug: visits of tocilizumab injection (every 4 weeks, up to 5 visits); Drug: Rituximab 375 mg/m2 at Day-30; Drug: Rituximab 375 mg/m2 at Day-15 (only for donors living); Other: Transplant Day-0
- Desensitization with Rituximab only (MFI<15000) (Other)
  Interventions: Drug: Rituximab 375 mg/m2 at Day-30; Drug: Rituximab 375 mg/m2 at Day-15 (only for donors living); Other: Transplant Day-0

INTERVENTIONS:
Drug: visits of tocilizumab injection (every 4 weeks, up to 5 visits) — every 4 weeks, up to 5 visits (D-170, D-142, D-114, D-86, D-58).
  Arms: Desensitization with Tocilizumab and rituximab (MFI >15000)
Drug: Rituximab 375 mg/m2 at Day-30 — Rituximab 375 mg/m2 at Day-30
Drug: Rituximab 375 mg/m2 at Day-15 (only for donors living) — Rituximab 375 mg/m2 at Day-15
Other: Transplant Day-0 — TRANSPLANTATION

SUMMARY:
Kidney transplantation is the best renal-replacement in the setting of end-stage renal disease. However, some transplant candidates have developed anti-HLA alloantibodies (human leukocyte antigen). When they are numerous and when their strength assessed by mean fluorescence intensity (MFI) is high it is very complicated to find-out a suitable kidney allograft against which the recipient has a negative cross-match. In such a case the only hope for the patient is desensitization therapy, whereby the treatment will decrease anti-HLA alloantibodies below a threshold, i.e. MFI < 3,000, enabling kidney transplantation without risking antibody-mediated rejection. Desensitization relies on i) apheresis technics in order to withdraw circulating anti-HLA antibodies, and ii) immunosuppression, i.e. rituximab or tocilizumab, targeting B-lymphocytes, and tacrolimus/mycophenolic acid/steroids targeting T-cells. The type of apheresis is guided by the pre-desensitization MFI of anti-HLA alloantibodies, e.g. double filtration plasmapheresis or semispecific immunoadsorption. Likely the choice between rituximab and tocilizumab depends also on predesensitization anti-HLA antibody MFIs. At the end of the desensitization process, the patient will be able to get a kidney transplant either from a live-donor or from a deceased donor.

ELIGIBILITY:
Inclusion Criteria:

* Patients on the kidney transplant list, waiting for a first or repeat transplant
* Presence of anti HLA antibodies either class I and/or II
* Sensitized against a potential living donor or have been on the waiting list for at least 3 years and having no potential live-donor
* Patients eligible for desensitization will receive either rituximab alone, or rituximab plus apheresis, or tocilizumab before rituximab
* Normal recent (<6 months) cardiac workup
* Vaccinated against pneumococcus and meningococcus B and C
* Willingness of the patient to undergo the desensitization process and Express consent of the patient
* for women of childbearing age, effective contraception or abstinence
* Affiliated to a social security scheme or of such a scheme

Exclusion Criteria:

* Active underlying infections or neoplasia
* Pregnant women, parturient or breastfeeding
* Subject in exclusion period of another study
* Subject under administrative or judicial control
* Subject who cannot be contacted in an emergency
* Rituximab contra indication: hypersensitivity (to active substance or murine protein), active and severe infections, patients in a severely immunocompromised state, severe heart failure or severe, uncontrolled cardiac disease.
* Tocilizumab contra indication: hypersensitivity, active and severe infections. Apheresis contra indication: active and severe infection, untreated or instable coagulation disorders, unstable coronary disease, recent stroke, hemodynamic instability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Description of the results of the strategy of desensitization in patients who will access to kidney transplantation from deceased or living donors. | at day 1 start of desensitization, at day 0 of Graft
  Decrease of MFI for highest donor-specific alloantibody (DSA) between start and end of desensitization for every patient in each category

SECONDARY OUTCOMES:
Desensitization efficacy with regards to DSA decrease and kidney transplantation | Day-198, at day-30 Graft, at day-15, at day0 of Graft,
  MFI for highest DSAs for each group
impairment of DSA synthesis | Day-198, at day-30 Graft, at day-15, at day0 of Graft,
  Decrease in peripheral plasma cells and plasmablasts of >50%
Impairment of immune response | Day-198, at day-30 Graft, at day-15, at day0 of Graft,
  Decrease in complement factors of >25%
Incidence of treatment desensitization protocols, emergent adverse events (safety and Tolerability) | Day-198, at day-30 Graft, at day-15
  Emergent adverse events to the desensitization therapy will be carefully monitored during the treatment period and within the following three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble Alpes University Hospital, La Tronche, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Orandi BJ, Montgomery RA, Segev DL. Kidney Transplants from HLA-Incompatible Live Donors and Survival. N Engl J Med. 2016 Jul 21;375(3):288-9. doi: 10.1056/NEJMc1604523. No abstract available. PMID 27468073
- [Result] Montgomery RA, Lonze BE, King KE, Kraus ES, Kucirka LM, Locke JE, Warren DS, Simpkins CE, Dagher NN, Singer AL, Zachary AA, Segev DL. Desensitization in HLA-incompatible kidney recipients and survival. N Engl J Med. 2011 Jul 28;365(4):318-26. doi: 10.1056/NEJMoa1012376. PMID 21793744
- [Result] Vo AA, Choi J, Cisneros K, Reinsmoen N, Haas M, Ge S, Toyoda M, Kahwaji J, Peng A, Villicana R, Jordan SC. Benefits of rituximab combined with intravenous immunoglobulin for desensitization in kidney transplant recipients. Transplantation. 2014 Aug 15;98(3):312-9. doi: 10.1097/TP.0000000000000064. PMID 24770617
- [Result] Kahwaji J, Jordan SC, Najjar R, Wongsaroj P, Choi J, Peng A, Villicana R, Vo A. Six-year outcomes in broadly HLA-sensitized living donor transplant recipients desensitized with intravenous immunoglobulin and rituximab. Transpl Int. 2016 Dec;29(12):1276-1285. doi: 10.1111/tri.12832. Epub 2016 Oct 24. PMID 27529314
- [Result] Klein K, Susal C, Schafer SM, Becker LE, Beimler J, Schwenger V, Zeier M, Schemmer P, Macher-Goeppinger S, Scherer S, Opelz G, Morath C. Living donor kidney transplantation in patients with donor-specific HLA antibodies enabled by anti-CD20 therapy and peritransplant apheresis. Atheroscler Suppl. 2013 Jan;14(1):199-202. doi: 10.1016/j.atherosclerosissup.2012.10.030. PMID 23357165
- [Result] Rostaing L, Maggioni S, Hecht C, Hermelin M, Faudel E, Kamar N, Sallusto F, Doumerc N, Allal A. Efficacy and safety of tandem hemodialysis and immunoadsorption to desensitize kidney transplant candidates. Exp Clin Transplant. 2015 Apr;13 Suppl 1:165-9. PMID 25894148
- [Result] Kauke T, Klimaschewski S, Schoenermarck U, Fischereder M, Dick A, Guba M, Stangl M, Werner J, Meiser B, Habicht A. Outcome after Desensitization in HLA or ABO-Incompatible Kidney Transplant Recipients: A Single Center Experience. PLoS One. 2016 Jan 5;11(1):e0146075. doi: 10.1371/journal.pone.0146075. eCollection 2016. PMID 26730981